CLINICAL TRIAL: NCT05064098
Title: Interpretations and Predictions of Patient Reported Outcomes by Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3576.cc
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-Surgical Breast Cancer Patients: Adult female patients newly diagnosed with stage 0-III breast cancer seen as a surgical consultation from 06/01/2019 to present.
- Breast Cancer Survivors: Breast Cancer Survivors

SUMMARY:
This study will assess how patients' long-term quality of life after different surgical approaches compares to their predicted quality of life.

DETAILED DESCRIPTION:
This study will assess how patients' long-term quality of life after different surgical approaches compares to their predicted quality of life. It will also provide the research team with improved understanding of how patients interact with and prefer to receive QOL information. Improved understanding of patient predictions and perceptions of information display will allow us to incorporate predicted future PROs into the shared decision making process as well as allow us to provide this important information to patients in a meaningful way.

ELIGIBILITY:
Inclusion Criteria:

* Pre-surgical female breast cancer patients
* Female breast cancer survivors

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pre-surgical breast cancer patients and breast cancer survivors
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Predicted patient reported outcomes up to 1 year after | 12 months
  Predicted patient reported outcomes for each domain six-months and 1 year after breast surgery.
Actual patient reported outcomes for each domain after surgery | 6 month
  Actual PRO scores for each domain six-months after surgery
Compare predicted and actual outcomes | 12 months
  Comparison of predicted versus actual PRO scores in patients undergoing surgery
Patients preferred method of communicating results | 12 months
  Patients' preferred means of receiving and communicating PRO results.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tevis, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hopspital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No